CLINICAL TRIAL: NCT00817622
Title: Effects of EPA Alone and Combined With Vitamin E on Blood Leptin, Adiponectin and Enzymatic Antioxidants Levels in Type II Diabetic Patients; A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effects of EPA and Vitamin E on Leptin, Adiponectin and Enzymatic Antioxidants in Type 2 DM
Acronym: EPA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Professor Mahmood Djalali, Tehran University of Medical Sciences
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 27-4955
Record Dates: First submitted 2009-01-03; First posted 2009-01-06 (Estimated); Last update posted 2009-11-18 (Estimated); Status verified 2009-11

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus type 2; EPA; leptin; adiponectin
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Placebo Comparator): Placebo, Placebo :
  Placebo pearls,500 mg QID for 12 Weeks (2000 mg corn oil per day) Placebo pearl + corn oil 400 mg per day for 12 weeks
  Interventions: Dietary Supplement: EPA, Vitamin E
- B (Active Comparator): EPA, Placebo :
  EPA pearls,500 mg QID for 12 Weeks (2000 mg per day),From MINAMINUTRITION Company(Belgium)+ Placebo pearl ,corn oil 400 mg per day for 12 weeks
  Interventions: Dietary Supplement: EPA, Vitamin E
- C (Placebo Comparator): Placebo ,Vitamin E :
  Placebo pearls,500 mg QID for 12 Weeks (2000 mg corn oil per day)+ Vitamin E pearls, 400 mg from DANA Company(IRAN) per day for 12 weeks
  Interventions: Dietary Supplement: EPA, Vitamin E
- D (Active Comparator): EPA, Vitamin E :
  EPA pearls,500 mg QID From MINAMINUTRITION Company(Belgium) for 12 Weeks (2000 mg EPA per day)+ Vitamin E pearls, 400 mg from DANA Company ( IRAN) per day for 12 weeks
  Interventions: Dietary Supplement: EPA, Vitamin E

INTERVENTIONS:
Dietary Supplement: EPA, Vitamin E — EPA pearls, 500 mg QID for 12 Weeks (2000 mg per day) Vitamin E pearls, 400 mg per day for 12 weeks
  Other Names: Plus EPA

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of EPA(Eicosapentaenoic Acid)alone and with VitE in diabetic patients.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo-controlled, parallel-group study design After a 12weeks, subjects with type II DM will be randomized to receive either 2000 mg pearl EPA per day plus a double-blinded matching placebo (1 corn oil pearls per day) for 12 weeks OR 400 mg VitE pearl plus double-blinded per day plus a double-blinded matching placebo (4 corn oil pearls per day) for 12 weeks OR 2000 mg pearl EPA per day plus a double-blinded matching 400 mg VitE pearl OR placebo(4corn oil pearls per day plus 1 corn oil pearls per day )for 12 weeks.The total dose of EPA pearl will be 2000 mg per day (with the EPA or matching placebo corn oil doses remaining at 4 pearls per day) and The total dose of VitE pearl will be 400 mg per day (with the VitE or matching placebo corn oil doses remaining at 1 pearls per day).

ELIGIBILITY:
Inclusion Criteria:

* DM Type II.
* Antidiabetic drug therapy which cannot be stopped.
* History of DM about 2-15 year.
* Age between 30-55 year.
* No History of circulatory, thyroid, pulmonary, liver, kidney, cancer.

Exclusion Criteria:

* DM Type I.
* Nephropathy.
* Retinopathy.
* Cancer.
* Thyroid disease.
* Renal failure.
* pulmonary disease
* MI.
* CHD.
* Liver disease,

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2007-01; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Changes in leptin and adiponectin after 12 Weeks | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mahmood Djalali, Professor, Study Chair — Tehran University of Medical Sciences, school of Public Health; Shokooh Sarbolouki, PhD Student, Principal Investigator — Tehran University of Medical Sciences, School of Public Health; Ahmad Reza - Dorosti, Ph.D., Study Chair — Tehran University of Medical Sciences,School of Public Health
Locations (1):
- Tehran University Of Medical Sciences, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Sarbolouki Sh, Djalali M, Dorosty A, Djazayery S, Eshraghian M, Ebadi S, Hashemi S. Effects of EPA and Vitamin E on Serum Enzymatic Antioxidants and Peroxidation Indices in Patients with Type II Diabetes Mellitus. Iran J Public Health. 2010;39(3):82-91. Epub 2010 Sep 30. PMID 23113026